CLINICAL TRIAL: NCT01792960
Title: Registry and Prevalence of Gene Mutation in Korean Patients With Familial Hypertrophic Cardiomyopathy
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2012-0869
Record Dates: First submitted 2013-02-07; First posted 2013-02-15 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Familial Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic, Familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — serum, whole blood, DNA
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- familial hypertrophic cardiomyopathy: familial hypertrophic cardiomyopathy patients and their relatives

SUMMARY:
Set the Korean Familial Hypertrophic Cardiomyopathy (KFHC) registry to study the prevalence of gene mutations in Korean patients with familial hypertrophic cardiomyopathy

ELIGIBILITY:
Inclusion Criteria:

1. left ventricular maximal wall thickness ≥ 15mm on echocardiography
2. hypertrophic cardiomyopathy patients' relatives

Exclusion Criteria:

1. other cardiomyopathy or systemic disease (e.g. fabry disease, danon disease, glycogen storage disease)
2. who deny the study entrance, especially in patients' relatives

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: familial hypertrophic cardiomyopathy patients and their relatives
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
1) DNA analysis | 1 year
  1) Identify susceptible genes for familial hypertrophic cardiomyopathy in Korean

SECONDARY OUTCOMES:
2) Prognosis of familial hypertrophic cariomyopathy | 1 year
  2) all-cause mortality, hospitalization for heart failure progression, stroke, heart transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital, Yonsei University College of Medicine, Seoul, Seoul, South Korea